CLINICAL TRIAL: NCT06137456
Title: First Report of a New Exoskeleton in Incomplete Spinal Cord Injury: FreeGait®
Brief Title: First Report of a New Exoskeleton in Incomplete Spinal Cord Injury
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara City Hospital Bilkent (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AnkaraCHBilkent-PMR-MSS-02
Record Dates: First submitted 2023-11-14; First posted 2023-11-18 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Spinal Cord Injuries; Walking, Difficulty
MeSH Terms: conditions — Spinal Cord Injuries; Mobility Limitation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study group (Experimental): Participants were involved in exoskeletal robotic therapy three days a week and conventional therapy five days a week for a maximum of eight weeks.
  Interventions: Device: Exoskeletal robotic therapy for walking.
- Control group (Active Comparator): Participants were involved in conventional therapy five days a week for a maximum of eight weeks.
  Interventions: Other: Conventional exercise therapy

INTERVENTIONS:
Device: Exoskeletal robotic therapy for walking. — Exoskeletal robotic therapy for walking. Therapy sessions were scheduled for 40 minutes each. The study group performed exoskeleton walking and balance exercises 3 days a week.
  Arms: Study group
Other: Conventional exercise therapy — Conventional treatment consisted of walking and balance exercises, stretching, strengthening, and mobility exercises, for 40 minutes, 5 days a week.
  Arms: Control group

SUMMARY:
The goal of this clinical trial is to compare the effects of exoskeletal robotic therapy and conventional exercise therapy in incomplete spinal cord injury (SCI). The main questions it aims to answer are:

* Is exoskeletal robotic therapy effective in improving functional ambulation in SCI?
* Is exoskeletal robotic therapy effective in enhancing Activities of Daily Living in SCI?

Participants treated with either:

* Exoskeletal robotic therapy along with conventional exercise therapy, or
* Only conventional exercise therapy.

DETAILED DESCRIPTION:
Background: Intensive walking practice is a task that requires performance above the limits of conventional therapy. As a solution, robot-assisted exoskeletons that allow walking on the ground are produced. The exoskeletons can allow the user to perform intense, targeted, and multi-repetitive movements and at the same time provide stability and balance during walking. In this study, a new robot-supported exoskeleton system was used for gait and balance rehabilitation. This study is important as the first clinical study of a new walking system. The primary aim of the study was to evaluate the effect of the FreeGait® exoskeleton system (BAMA Technology, Ankara, Türkiye) on gait parameters in patients with motor incomplete spinal cord injury. The secondary aim was to assess its impact on quality of life and independence.

Methods: Fourteen participants with incomplete spinal cord injury were included in the study. An average of 20.7 sessions of exoskeleton therapy was administered to the study group. Gait training was attempted to be diversified as much as possible during the exoskeleton training. 10MWT, Timed Up and Go Test (TUG), WISCI II, Berg Balance Scale (BBS), Visual Analogue Scale (VAS) for fear of falling, Spinal Cord Independence Measure (SCIM III), World Health Organization Quality of Life Scale-Short Form (WHOQOL - BREF) were used for evaluation.

Results: WISCI II levels improved significantly in the study group (p = 0.031). Overground walking speed means calculated from 10MWT increased by 66%, twofold compared to the control group (p = 0.016, p = 0.063, respectively). The mobility subscale of SCIM III, the total SCIM III scores, and the WHOQOL-BREF physical health domain score increased significantly, contrary to the control group (p < 0.05). However, there was no difference in the mean change of all measurements between groups (p > 0.05).

Conclusions: Gait training with the new exoskeleton system contributes to functional walking skills. It is possible that the residual motor learning ability, together with the balance and compensation mechanisms, played a role in the outcome. It is also important that this improvement in functional mobility is reflected in ADLs. It can be supposed that walking in different patterns, and speeds gives a way to simulate daily living conditions, which is the basis of the achievements in this study.

ELIGIBILITY:
Inclusion Criteria:

* SCI below T4,
* Patients with AIS (American Spinal Injury Association Impairment Scale) C or D injury,
* Bilateral quadriceps femoris manual test scores ≥ 2,
* Upper extremity manual muscle test scores = 5,
* Participants with adequate spinal stabilization

Exclusion Criteria:

* Severe spasticity (Modified Ashworth Scale ≥ 3),
* Difference in leg length,
* Pregnancy, osteoporosis,
* Contracture, or limited range of motion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2023-11-01 (Actual); Study Completion 2023-11-01 (Actual)

PRIMARY OUTCOMES:
Walking Index in Spinal Cord Injury II | 23 months
  Walking Index in Spinal Cord Injury II for walking independence level assessment

SECONDARY OUTCOMES:
Ten-Meter Walking Test | 23 months
  Ten-Meter Walking Test for overground walking speed assessment
Timed Up and Go Test | 23 months
  Timed Up and Go Test overground walking assessment
Berg Balance Scale | 23 months
  Berg Balance Scale for balance assessment
Visual Analogue Scale | 23 months
  Visual Analogue Scale (VAS) for fear of falling assessment
Spinal Cord Independence Measure (SCIM III) | 23 months
  Spinal Cord Independence Measure (SCIM III) for activity of daily living assessment
World Health Organization Quality of Life Scale-Short Form (WHOQOL - BREF) | 23 months
  World Health Organization Quality of Life Scale-Short Form (WHOQOL - BREF) for quality of life assessment

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara City Hospital, Ankara, Turkey (Türkiye)

REFERENCES:
- [Background] Finlayson ML, Peterson EW. Falls, aging, and disability. Phys Med Rehabil Clin N Am. 2010 May;21(2):357-73. doi: 10.1016/j.pmr.2009.12.003. PMID 20494282
- [Background] Contreras-Vidal JL, A Bhagat N, Brantley J, Cruz-Garza JG, He Y, Manley Q, Nakagome S, Nathan K, Tan SH, Zhu F, Pons JL. Powered exoskeletons for bipedal locomotion after spinal cord injury. J Neural Eng. 2016 Jun;13(3):031001. doi: 10.1088/1741-2560/13/3/031001. Epub 2016 Apr 11. PMID 27064508
- [Background] Esquenazi A, Talaty M, Packel A, Saulino M. The ReWalk powered exoskeleton to restore ambulatory function to individuals with thoracic-level motor-complete spinal cord injury. Am J Phys Med Rehabil. 2012 Nov;91(11):911-21. doi: 10.1097/PHM.0b013e318269d9a3. PMID 23085703
- [Background] Fouad K, Tetzlaff W. Rehabilitative training and plasticity following spinal cord injury. Exp Neurol. 2012 May;235(1):91-9. doi: 10.1016/j.expneurol.2011.02.009. Epub 2011 Feb 17. PMID 21333646
- [Background] Leech KA, Kinnaird CR, Holleran CL, Kahn J, Hornby TG. Effects of Locomotor Exercise Intensity on Gait Performance in Individuals With Incomplete Spinal Cord Injury. Phys Ther. 2016 Dec;96(12):1919-1929. doi: 10.2522/ptj.20150646. Epub 2016 Jun 16. PMID 27313241
- [Background] Barbeau H, Norman K, Fung J, Visintin M, Ladouceur M. Does neurorehabilitation play a role in the recovery of walking in neurological populations? Ann N Y Acad Sci. 1998 Nov 16;860:377-92. doi: 10.1111/j.1749-6632.1998.tb09063.x. PMID 9928326
- [Background] Dobkin B, Barbeau H, Deforge D, Ditunno J, Elashoff R, Apple D, Basso M, Behrman A, Harkema S, Saulino M, Scott M; Spinal Cord Injury Locomotor Trial Group. The evolution of walking-related outcomes over the first 12 weeks of rehabilitation for incomplete traumatic spinal cord injury: the multicenter randomized Spinal Cord Injury Locomotor Trial. Neurorehabil Neural Repair. 2007 Jan-Feb;21(1):25-35. doi: 10.1177/1545968306295556. PMID 17172551
- [Background] Yang JF, Musselman KE, Livingstone D, Brunton K, Hendricks G, Hill D, Gorassini M. Repetitive mass practice or focused precise practice for retraining walking after incomplete spinal cord injury? A pilot randomized clinical trial. Neurorehabil Neural Repair. 2014 May;28(4):314-24. doi: 10.1177/1545968313508473. Epub 2013 Nov 8. PMID 24213960
- [Background] Colombo G, Wirz M, Dietz V. Driven gait orthosis for improvement of locomotor training in paraplegic patients. Spinal Cord. 2001 May;39(5):252-5. doi: 10.1038/sj.sc.3101154. PMID 11438840
- [Background] Hesse S, Uhlenbrock D. A mechanized gait trainer for restoration of gait. J Rehabil Res Dev. 2000 Nov-Dec;37(6):701-8. PMID 11321006
- [Background] Hesse S. Treadmill training with partial body weight support after stroke: a review. NeuroRehabilitation. 2008;23(1):55-65. PMID 18356589
- [Background] Calabro RS, Cacciola A, Berte F, Manuli A, Leo A, Bramanti A, Naro A, Milardi D, Bramanti P. Robotic gait rehabilitation and substitution devices in neurological disorders: where are we now? Neurol Sci. 2016 Apr;37(4):503-14. doi: 10.1007/s10072-016-2474-4. Epub 2016 Jan 18. PMID 26781943
- [Background] Esquenazi A, Talaty M, Jayaraman A. Powered Exoskeletons for Walking Assistance in Persons with Central Nervous System Injuries: A Narrative Review. PM R. 2017 Jan;9(1):46-62. doi: 10.1016/j.pmrj.2016.07.534. Epub 2016 Aug 24. PMID 27565639
- [Background] Bolliger M, Blight AR, Field-Fote EC, Musselman K, Rossignol S, Barthelemy D, Bouyer L, Popovic MR, Schwab JM, Boninger ML, Tansey KE, Scivoletto G, Kleitman N, Jones LAT, Gagnon DH, Nadeau S, Haupt D, Awai L, Easthope CS, Zorner B, Rupp R, Lammertse D, Curt A, Steeves J. Lower extremity outcome measures: considerations for clinical trials in spinal cord injury. Spinal Cord. 2018 Jul;56(7):628-642. doi: 10.1038/s41393-018-0097-8. Epub 2018 Apr 27. PMID 29700477
- [Background] Jackson AB, Carnel CT, Ditunno JF, Read MS, Boninger ML, Schmeler MR, Williams SR, Donovan WH; Gait and Ambulation Subcommittee. Outcome measures for gait and ambulation in the spinal cord injury population. J Spinal Cord Med. 2008;31(5):487-99. doi: 10.1080/10790268.2008.11753644. PMID 19086706
- [Background] Ditunno JF Jr, Ditunno PL, Scivoletto G, Patrick M, Dijkers M, Barbeau H, Burns AS, Marino RJ, Schmidt-Read M. The Walking Index for Spinal Cord Injury (WISCI/WISCI II): nature, metric properties, use and misuse. Spinal Cord. 2013 May;51(5):346-55. doi: 10.1038/sc.2013.9. Epub 2013 Mar 5. PMID 23459122
- [Background] Sahin F, Yilmaz F, Ozmaden A, Kotevolu N, Sahin T, Kuran B. Reliability and validity of the Turkish version of the Berg Balance Scale. J Geriatr Phys Ther. 2008;31(1):32-7. doi: 10.1519/00139143-200831010-00006. PMID 18489806
- [Background] Wirz M, Muller R, Bastiaenen C. Falls in persons with spinal cord injury: validity and reliability of the Berg Balance Scale. Neurorehabil Neural Repair. 2010 Jan;24(1):70-7. doi: 10.1177/1545968309341059. Epub 2009 Aug 12. PMID 19675123
- [Background] Unalan H, Misirlioglu TO, Erhan B, Akyuz M, Gunduz B, Irgi E, Arslan HE, Baltaci A, Aslan S, Palamar D, Kutlu A, Majlesi J, Akarirmak U, Karamehmetoglu SS. Validity and reliability study of the Turkish version of Spinal Cord Independence Measure-III. Spinal Cord. 2015 Jun;53(6):455-60. doi: 10.1038/sc.2014.249. Epub 2015 Feb 10. PMID 25665539
- [Background] Itzkovich M, Gelernter I, Biering-Sorensen F, Weeks C, Laramee MT, Craven BC, Tonack M, Hitzig SL, Glaser E, Zeilig G, Aito S, Scivoletto G, Mecci M, Chadwick RJ, El Masry WS, Osman A, Glass CA, Silva P, Soni BM, Gardner BP, Savic G, Bergstrom EM, Bluvshtein V, Ronen J, Catz A. The Spinal Cord Independence Measure (SCIM) version III: reliability and validity in a multi-center international study. Disabil Rehabil. 2007 Dec 30;29(24):1926-33. doi: 10.1080/09638280601046302. Epub 2007 Mar 5. PMID 17852230
- [Background] Development of the World Health Organization WHOQOL-BREF quality of life assessment. The WHOQOL Group. Psychol Med. 1998 May;28(3):551-8. doi: 10.1017/s0033291798006667. PMID 9626712
- [Background] Spampinato D, Celnik P. Multiple Motor Learning Processes in Humans: Defining Their Neurophysiological Bases. Neuroscientist. 2021 Jun;27(3):246-267. doi: 10.1177/1073858420939552. Epub 2020 Jul 25. PMID 32713291
- [Background] Li Y, Hollis ER 2nd. The role of motor network reorganization during rehabilitation. Neural Regen Res. 2017 May;12(5):745-746. doi: 10.4103/1673-5374.206641. No abstract available. PMID 28616027
- [Background] Wirz M, van Hedel HJA. Balance, gait, and falls in spinal cord injury. Handb Clin Neurol. 2018;159:367-384. doi: 10.1016/B978-0-444-63916-5.00024-0. PMID 30482328
- [Background] Gorgey AS. Robotic exoskeletons: The current pros and cons. World J Orthop. 2018 Sep 18;9(9):112-119. doi: 10.5312/wjo.v9.i9.112. eCollection 2018 Sep 18. PMID 30254967
- [Background] Laut J, Porfiri M, Raghavan P. The Present and Future of Robotic Technology in Rehabilitation. Curr Phys Med Rehabil Rep. 2016 Dec;4(4):312-319. doi: 10.1007/s40141-016-0139-0. Epub 2016 Nov 19. PMID 28603663
- [Background] van Hedel HJ; EMSCI Study Group. Gait speed in relation to categories of functional ambulation after spinal cord injury. Neurorehabil Neural Repair. 2009 May;23(4):343-50. doi: 10.1177/1545968308324224. Epub 2008 Nov 25. PMID 19036717
- [Background] Baunsgaard CB, Nissen UV, Brust AK, Frotzler A, Ribeill C, Kalke YB, Leon N, Gomez B, Samuelsson K, Antepohl W, Holmstrom U, Marklund N, Glott T, Opheim A, Penalva JB, Murillo N, Nachtegaal J, Faber W, Biering-Sorensen F. Exoskeleton gait training after spinal cord injury: An exploratory study on secondary health conditions. J Rehabil Med. 2018 Sep 28;50(9):806-813. doi: 10.2340/16501977-2372. PMID 30183055
- [Background] Wright MA, Herzog F, Mas-Vinyals A, Carnicero-Carmona A, Lobo-Prat J, Hensel C, Franz S, Weidner N, Vidal J, Opisso E, Rupp R. Multicentric investigation on the safety, feasibility and usability of the ABLE lower-limb robotic exoskeleton for individuals with spinal cord injury: a framework towards the standardisation of clinical evaluations. J Neuroeng Rehabil. 2023 Apr 12;20(1):45. doi: 10.1186/s12984-023-01165-0. PMID 37046307
- [Background] de Franca IS, Coura AS, de Franca EG, Basilio NN, Souto RQ. [Quality of life of adults with spinal cord injury: a study using the WHOQOL-bref]. Rev Esc Enferm USP. 2011 Dec;45(6):1364-71. doi: 10.1590/s0080-62342011000600013. Portuguese. PMID 22241194
- [Background] Ahuja CS, Wilson JR, Nori S, Kotter MRN, Druschel C, Curt A, Fehlings MG. Traumatic spinal cord injury. Nat Rev Dis Primers. 2017 Apr 27;3:17018. doi: 10.1038/nrdp.2017.18. PMID 28447605
- [Derived] Sipal MS, Yasar E, Ozisler Z, Adiguzel E, Yildirim S, Deler O, Kirdis S, Celik HI, Ulusahin SB, Kayalar G, Karaduman AA. First report of a new exoskeleton in incomplete spinal cord injury: FreeGait(R). J Spinal Cord Med. 2026 Jan;49(1):118-128. doi: 10.1080/10790268.2024.2426314. Epub 2024 Nov 22. PMID 39576286